CLINICAL TRIAL: NCT06875986
Title: REXULTI Drug General Use-results Survey (Excessive Motor Activity or Physically/Verbally Aggressive Behavior Due to Rapid Changes in Mood, Irritability, and/or Outbursts Associated With Dementia Due to Alzheimer's Disease)
Status: Recruiting | Type: Observational
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 331-101-00612
Record Dates: First submitted 2025-03-12; First posted 2025-03-14 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — brexpiprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Brexpiprazole (Rexulti) — In general, for adults, start with taking 0.5 mg of brexpirazole at a time, once a day. Then the dose will be increased with an interval of at least one week to 1 mg at a time, once a day. If you have no problem with tolerability and do not show an adequate response, the dose may be increased to 2 mg at a time, once a day, but the increase should be made at intervals of at least one week.

SUMMARY:
The purpose of this study is to evaluate safety of REXULTI in patients under daily clinical settings. In addition, information on efficacy will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Alzheimer's disease

Exclusion Criteria:

-

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in Japan who are planned to be newly started on Brexpiprazole OD tablets therapy for the excessive motor activity or physically/verbally aggressive behavior due to rapid changes in mood, irritability, and/or outbursts associated with dementia due to Alzheimer's disease
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-23 (Estimated)

PRIMARY OUTCOMES:
Safety Information (Adverse Event) | 24 weeks from the initiation of brexpiprazole treatment
  Any untoward medicinal occurrence in a patient or clinical study subject administered a Medicinal Product and which does not necessarily have a causal relationship with this treatment (ICH-E2A Guideline). An Adverse Event can therefore be any unfavorable and unintended sign (e.g. abnormal laboratory finding), symptom, or disease temporally associated with the use of a Medicinal Product (brexpiprazole), whether or not it is considered causally related to the Medicinal Product.
Safety Information (Special Situations) | 24 weeks from the initiation of brexpiprazole treatment
  Situations related to the use of an Otsuka product which may or may not be associated with an adverse event: -Maternal (pregnancy and breastfeeding) or paternal (via semen) exposure; -Exposure during breastfeeding; -Overdose/Incorrect dosage, misuse, abuse (e.g. patient sharing products); -Medication errors (e.g. patient took wrong dose); -Lack of therapeutic efficacy (e.g. the product doesn't work); -Occupational exposure (e.g.: nurse administering the product is exposed); -Cases of suspected transmission of infectious agents; -Use of suspected or confirmed falsified product(s) or quality defect of the product(s); -Withdrawal reactions; -Accidental exposure (e.g.: child takes parent's product); -Drug-drug/drug-food interactions; -Unintentional use of product in a non-approved population (e.g.: pediatric or geriatric population); -Disease progression/exacerbation of existing disease
Safety Information (Number of off-Label Use) | 24 weeks from the initiation of brexpiprazole treatment
  Collecting any type of off-Label Use that refers to situations where a product is intentionally used for a medical purpose not in accordance with the authorized product information. Off-label use also includes the intentional use in non-authorized population categories not indicated in the label.
Safety Information (Serious Adverse Event) | 24 weeks from the initiation of brexpiprazole treatment
  Any adverse drug experience/event occurring at any dose which -results in death -is life-threatening -requires inpatient hospitalization or prolonged of existing hospitalization -results in persistent or significant disability or incapacity -is a congenital anomaly/birth defect -is medically significant.
Safety Information (Non-serious Adverse Events) | 24 weeks from the initiation of brexpiprazole treatment
  All Adverse Events that do not meet the definition of a serious Adverse Event are considered non-serious Adverse Events.

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmacovigilance Department, Osaka, Osaka, Japan